CLINICAL TRIAL: NCT02972216
Title: A Post-marketing Surveillance Study to Evaluate the Effectiveness and Safety of Docetaxel-Based Chemotherapy
Brief Title: Post-marketing Surveillance Study of Docetaxel-Based Chemotherapy
Status: Completed | Type: Observational
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YSP RFH3001-01
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Nonsmall Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Nolbaxol: For Nonsmall Cell Lung Cancer (NSCLC) Docetaxel (either Group I or Group II) 60 mg/m2 will be administrated by intravenous infusion for 1 hour every 3 weeks (a study medication cycle) and up to 4 study medication cycles throughout this study. For Squamous Cell Carcinoma of the Head and Neck (SCCHN) Docetaxel (either Group I or Group II) 60 mg/m2 will be administrated by intravenous infusion for 1 hour followed by cisplatin 60 ~ 75 mg/m2 for 1-3 hours or based on the general practice of the site every 3 weeks and up to 4 study medication cycles throughout this study.
  Interventions: Drug: Nolbaxol; Drug: cisplatin
- Taxotere: For Nonsmall Cell Lung Cancer (NSCLC) Docetaxel (either Group I or Group II) 60 mg/m2 will be administrated by intravenous infusion for 1 hour every 3 weeks (a study medication cycle) and up to 4 study medication cycles throughout this study. For Squamous Cell Carcinoma of the Head and Neck (SCCHN) Docetaxel (either Group I or Group II) 60 mg/m2 will be administrated by intravenous infusion for 1 hour followed by cisplatin 60 ~ 75 mg/m2 for 1-3 hours or based on the general practice of the site every 3 weeks and up to 4 study medication cycles throughout this study.
  Interventions: Drug: Taxotere; Drug: cisplatin

INTERVENTIONS:
Drug: Nolbaxol
  Other Names: docetaxel
  Groups: Nolbaxol
Drug: Taxotere
  Other Names: docetaxel
  Groups: Taxotere
Drug: cisplatin

SUMMARY:
A Post-marketing Surveillance Study to Evaluate the Effectiveness and Safety of Docetaxel-Based Chemotherapy

ELIGIBILITY:
Inclusion Criteria:

-Histologically or cytologically confirmed unresectable locally advanced NSCLC with progressed or recurred after no more than four previous docetaxel-free chemotherapy regimens, or unresectable locally advanced or metastatic SCCHN or recurred after previous docetaxel-free chemotherapy regimens

Exclusion Criteria:

1. Women who are nursing or pregnant during the study period;
2. Patients with carcinoid tumors, small-cell carcinoma of the lung;
3. A history of another malignancy within the last five years (except for cured basal cell carcinoma of the skin and cured carcinoma in situ of the uterine cervix);
4. Any other morbidity or situation with contraindications for chemotherapy (e.g. active infection, myocardial infarction in the preceding 6 months);
5. Neutrophil counts < 1,500 cells/mm3;
6. A history of hypersensitivity to docetaxel or cisplatin;
7. Symptomatic heart disease including unstable angina, congestive heart failure or uncontrolled arrhythmias;
8. Subjects have active hepatitis;
9. Subjects are known positive for Human Immunodeficiency Virus (HIV);
10. Any condition judged by investigator, participates the study will jeopardize patient's wellbeing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 40 evaluable patients with locally advanced or metastatic NSCLC, SCCHN or esophageal cancer will be equally randomized to either Nolbaxol or Taxotere.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Every 8 weeks after post-dosing follow-up visit, and conducted until disease progression or up to 11 months.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Every 8 weeks after post-dosing follow-up visit, and conducted until disease progression or up to 11 months.
Adverse Events as a measure on safety | Adverse event will be evaluated during the study regimens treatment period and up to 8 weeks after the last dose of study regimen visit.